CLINICAL TRIAL: NCT06489184
Title: This is a Multicenter, Retrospective Real-world Study of Zanubrutinib in the Treatment of Chronic Lymphocytic Leukemia in China
Brief Title: The Real World Study of Zanubrutinib in the Treatment of Chronic Lymphocytic Leukemia in China
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Other Study IDs: 2024Zanu-RW-01
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: CLL
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Zanubrutinib — patients with treatment naive or R/R CLL who treatment with Zanubrutinib

SUMMARY:
This is a Multicenter, Retrospective Real-world Study of Zanubrutinib in the Treatment of Chronic Lymphocytic Leukemia in China

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged ≥18 years old
* 2. Must have a confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL) requiring treatment (iwCLL [International Workshop on Chronic Lymphocytic Leukemia] criteria)；
* 3. Treatment-naïve OR Refractory Recurrence CLL patients who were initiated on Zanubrutinib;
* 4.Prior or current use of Zanubrutinib for ≥3 months
* 5.At least one follow-up was recorded during Zanubrutinib treatment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators participating in this observational study should include all patients with CLL who initiated treatment with zanubrutinib over the period from July 1st, 2020 to the present, regardless of the treatment status at the time of inclusion. Thus, at the time of enrolment and retrospective data collection, patients may still be on treatment or have stopped treatment for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to two years
  PFS is defined as the duration from date of Zanubrutinib initiation to date of disease progression (PD [according to the physician's evaluation]) or death from any cause

SECONDARY OUTCOMES:
Overall Survival | up to two years
  OS is defined as the time from the starting date of Zanubrutinib to the date of death due to any cause.
Time to Next Therapy (TTNT) | up to two years
  The TTNT will be calculated as the difference between Zanubrutinib initiation date and initiation date of the first next therapy for CLL
Adverse Events | up to two years
  Percentage of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Special Situations

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided